CLINICAL TRIAL: NCT04721197
Title: Program Evaluation: Eggs Hatching Hope. Providing Egg Vouchers to Women With Young Children in Rural Honduras.
Brief Title: Hens Hatching Hope
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Southern University (Other)
Collaborators: Shoulder to Shoulder (Other)
Responsible Party: Principal Investigator, Ana Palacios, Assistant Professor, Georgia Southern University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2012965659
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Malnutrition, Child
Keywords: Stunting; Eggs; diarrhea; complementary foods
MeSH Terms: conditions — Child Nutrition Disorders; Growth Disorders; Diarrhea | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The principal investigator and statistician will be blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 30-day egg vouchers, in addition to the standard of care.
  Interventions: Other: Egg vouchers; Other: Standard of Care
- Control group (Active Comparator): Standard of care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Egg vouchers — 30-day egg vouchers will be provided monthly, in addition to standard of care.
  Arms: Intervention
Other: Standard of Care — Participants will continue to receive the standard of care. No egg vouchers.

SUMMARY:
The study is a prospective community-cluster non-randomized trial that will evaluate the effectiveness of a program that will provide 30-day egg vouchers to mothers of 6 to 24 month-old children living in rural areas of Intibucá, Honduras.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children ages 6 to 24 months at the time the study begins
* No cerebral palsy, birth defect or condition that may affect their growth or development.
* Children living in the department of Intibucá, Honduras

Exclusion Criteria:

* Children from families that are considering leaving the region within the next 12 months
* Known egg allergy

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2021-01-23 (Actual); Primary Completion 2026-01-22 (Estimated); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
Changes in Length/Height-for-age z-scores (zHAZ) from baseline at 6 months | 6 months
  Calculated using the 2006 World Health Organization Child Growth Standards
Changes in Length/Height-for-age z-scores (zHAZ) from baseline at 12 months | Change from baseline zHAZ at 12 months
  Calculated using the 2006 World Health Organization Child Growth Standards

SECONDARY OUTCOMES:
Changes in the prevalence of stunting from baseline at 6 months | 6 months
  Calculated using the 2006 World Health Organization Child Growth Standards (zHAZ <-2)
Changes in the prevalence of stunting from baseline at 12 months | 12 months
  Calculated using the 2006 World Health Organization Child Growth Standards (zHAZ <-2)
Changes in the prelavence of underweight (Weight-for-age z-score <-2) from baseline at 6 months | 6 months
  Calculated using the 2006 World Health Organization Child Growth Standards
Changes in the prelavence of underweight (Weight-for-age z-score <-2) from baseline at 12 months | 12 months
  Calculated using the 2006 World Health Organization Child Growth Standards
Assessment of rapid weight gain after 6 months of intervention | 6 months
  Defined as a zBMI upward percentile crossing (>+0.67 SD) Calculated using the 2006 World Health Organization Child Growth Standards
Assessment of rapid weight gain after 12 months of intervention | 12 months
  Defined as a zBMI upward percentile crossing (>+0.67 SD) Calculated using the 2006 World Health Organization Child Growth Standards
Changes in the prevalence of diarrhea from baseline at 12 months | 12 months
  Defined as three or more liquid or semisolid stools in 24 hours
Changes in the prevalence of Respiratory symptoms from baseline at 12 months | 12 months
  Defined as reported presence of cough, or nasal congestion, or ear ache, or sore throat in the last 7 days.
Changes in the prevalence of Respiratory infections from baseline at 12 months | baseline and 12 months
  Defined as reported presence of fever + any of the following symptoms: cough, or nasal congestion, or ear ache, or sore throat in the last 7 days
Changes in the food insecurity scores from baseline at 6 months | 6 months
  Measured using the 2012 Latin American and Caribbean scale of Food insecurity (Escala Latinoamercana y Caribeña de Seguridad Alimentaria)
Changes in the food insecurity scores from baseline at 12 months | 12 months
  Measured using the 2012 Latin American and Caribbean scale of Food insecurity (Escala Latinoamercana y Caribeña de Seguridad Alimentaria)
Changes in the dietary diversity scores from baseline at 6 months | 6 months
  Measured using the frequency of intake survey from the 2012 Latin American and Caribbean scale of Food insecurity (Escala Latinoamercana y Caribeña de Seguridad Alimentaria)
Changes in the dietary diversity scores from baseline at 12 months | 12 months
  Measured using the frequency of intake survey from the 2012 Latin American and Caribbean scale of Food insecurity (Escala Latinoamercana y Caribeña de Seguridad Alimentaria)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Palacios, MD, PhD, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Clinica medica Roy and Melaney Sanders, Concepción, Intibucá Department, Honduras